CLINICAL TRIAL: NCT02640885
Title: Use of Foley's Catheter Balloon Tamponade to Control Placental Site Bleeding Resulting From Placenta Previa During Cesarean Section
Brief Title: The Foley's Catheter Balloon to the Bleeding From Placenta Previa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCB
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Foley's cather tamponade (Experimental): Balloon tamponade with 2-way Foley's Cather was successfully used during cesarean section due to sever postpartum haemorrhage after failure of medical treatment.
  Interventions: Device: Foley's cather ballon

INTERVENTIONS:
Device: Foley's cather ballon

SUMMARY:
Post-partum haemorrhage due to placenta previa is usually from the placental bed at the lower uterine segment and it occurs after the placenta separation. Although, nowadays the obstetrician can diagnose placenta previa before delivery, it is still one of the important causes of maternal mortality . Hysterectomy can be the only effective action to take, although it carries many morbidities for the women especially those with low parity.

Uterine packing considers as a line of treatment before performing surgical procedures in postpartum hemorrhage resulting from placental site bleeding. It can save life, avoid laparotomy and save uterus.

Nowadays, the use of intrauterine balloons have been developed and become effective for the control of placental site bleeding not responding to medical treatment. The 2-way Foley's Cather has many advantages over the gauze packing; First, it allows drainage of blood so no occult bleeding could be accumulated inside the uterus as in uterine gauze, second the removal of the Foley's Cather balloon is easy and not a painful, third, the removal of 2-way Foley's Cather could be gradually as a test of its effectiveness before complete removal .

ELIGIBILITY:
Inclusion Criteria:

* Patients with placenta previa
* Delivered by cesarean section

Exclusion Criteria:

* Patients with sever uncontrolled uterine bleeding after delivery
* Placenta accreta

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Amount of blood loss (mL) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided